CLINICAL TRIAL: NCT05963009
Title: Randomized, Open Label, Crossover Study to Evaluate the Relative Bioavailability of a New Tablet Formulation of CIN-107 as Compared to Oral Solution and to Assess the Effect of Food on the CIN-107 Tablet Formulation in Healthy Subjects
Brief Title: Baxdrostat Bioavailability and Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-112
Record Dates: First submitted 2023-07-03; First posted 2023-07-27 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: pharmacokinetics (PK); food effect; bioavailability
MeSH Terms: conditions — Hypertension | interventions — Solutions; Tablets

STUDY DESIGN:
Intervention Model Description: Randomized Crossover between 1) oral solution, 2) tablet in the fasted state, and 3) tablet in the fed state
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Baxdrostat oral solution (Experimental): 5 mg CIN-107 oral solution in a fasted state
  Interventions: Drug: baxdrostat (formerly CIN-107) oral solution
- Baxdrostat tablet (fasted state) (Experimental): 5 mg CIN-107 tablet(s) in a fasted state
  Interventions: Drug: baxdrostat (formerly CIN-107) oral solution
- Baxdrostat tablet (fed state) (Experimental): 5 mg CIN-107 tablet(s) in a fed state (standard high fat meal)
  Interventions: Drug: baxdrostat (formerly CIN-107) oral solution

INTERVENTIONS:
Drug: baxdrostat (formerly CIN-107) oral solution — 5 mg single dose of baxdrostat given as either a solution or tablet in either the fed or fasted state, depending on the arm of the study
  Other Names: baxdrostat (formerly CIN-107) tablet

SUMMARY:
The goal of this study was to compare the characteristics of a new tablet formulation versus an oral solution of CIN-107 (baxdrostat) in terms of CIN-107 levels over time in the blood and to compare the effect of food on these parameters in healthy volunteer participants who received the CIN-107 tablet under fed versus fasted conditions.

DETAILED DESCRIPTION:
The goals of this study were to:

1. To assess the safety and tolerability of single doses of CIN-107 tablet and oral solution in healthy participants.
2. Compare CIN-107 levels over time in the blood in participants after dosing between a tablet formulation of CIN-107 as compared to the oral solution.
3. Compare the CIN-107 levels over time in the blood in participants following dosing with a CIN-107 tablet after a meal versus in the fasted state.

Participants took either the oral solution or a tablet of CIN-107 and had their safety and blood levels of CIN-107 measured over several days following administration of CIN-107 tablet either in the fasted state or after a meal. The CIN-107 blood levels over time were compared between the groups given either the oral solution or the tablet and between the group given the CIN-107 tablet with a meal versus in the fasted state.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 55 years, inclusive, in good health based on medical and psychiatric history, physical examination, electrocardiogram (ECG), vital signs (seated and orthostatic), and routine laboratory tests (blood chemistry, hematology, coagulation, and urinalysis).
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive.
3. Nonsmokers who have not used nicotine-containing products for at least 6 months prior to Screening.
4. Male subjects with female partners of child-bearing potential must agree to use two medically accepted, highly effective methods of birth control from Day 1 through 90 days after the final dose of study drug.
5. Male subjects must agree to abstain from sperm donation from Day 1 through 90 days after administration of the final dose of study drug.
6. Female subjects with male partners must be surgically sterile (hysterectomy and/or bilateral oophorectomy), postmenopausal for at least 1 year (with follicle-stimulating hormone in postmenopausal range), or agree to use two medically accepted, highly effective methods of birth control from Day -14 until 60 days following the final dose of study drug.
7. Able to understand and willing to comply with study procedures and restrictions (including confinement to the clinical unit, fasting and meal requirements, and restrictions on physical activity, use of recreational drugs or alcohol, and medications), and provide written informed consent according to institutional and regulatory guidelines.

Exclusion Criteria:

1. Actively participating in an experimental therapy study; received experimental therapy with a small molecule other than CIN-107 within 30 days of the first dose of study drug, or 5 halflives, whichever is longer; or received experimental therapy with a large molecule within 90 days of the first dose of study drug, or 5 half-lives, whichever is longer.
2. A personal or family history of long QT syndrome, Torsades de Pointes, or other complex ventricular arrhythmias, or family history of sudden death.
3. History of, or current, clinically significant arrhythmias as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, atrial fibrillation, sinus node dysfunction, or clinically significant heart block. Subjects with minor forms of ectopy (eg, premature atrial contractions) are not necessarily excluded.
4. Prolonged QTcF (>450 msec).
5. Seated blood pressure higher than 150/90 mmHg or lower than 90/50.
6. Resting heart rate higher than 100 bpm or lower than 50 bpm.
7. Temperature (T) greater than 37.6 C (99.68 F), measured orally, and respiration rate less than 12 or greater than 20 breaths/minute.
8. Postural tachycardia (i.e. >30 bpm upon standing) or orthostatic hypotension (i.e., a fall in systolic blood pressure (SBP) of ≥20 mm Hg or diastolic blood pressure (DBP) of ≥ 10 mm Hg when a person assumes a standing position).
9. Serum potassium > upper limit of normal of the reference range (ULN) and serum sodium < lower limit of normal of the reference range (LLN).
10. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) values > 1.2 ULN.
11. Positive for human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody, or Hepatitis B surface antigen (HBsAg).
12. Any other clinical laboratory values which are meaningfully outside of normal limits (based on laboratory normal range) in the opinion of the Investigator.
13. A known history of porphyria, myopathy, or an active liver disease.
14. Evidence or history of any clinically significant immunologic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, musculoskeletal, hepatic, psychiatric, neurologic, or allergic disease (including clinically significant or multiple drug allergies); surgical conditions; cancer (with the exception of basal or squamous cell carcinoma of the skin and cancer that resolved or has been in remission for >5 years prior to Screening); or any condition that, in the Investigator's opinion, may confound study procedures or results, impact subject safety, or interfere with the absorption, distribution, metabolism, or excretion of the study drug (appendectomy allowed, cholecystectomy prohibited).
15. Use of any prescription medications (including topicals) or over-the-counter medications (other than occasional use of acetaminophen or nonsteroidal anti-inflammatory drugs, such as ibuprofen or naproxen, according to the package insert); herbal supplements; dietary supplements; or nutraceuticals within 14 days prior to the first dose of study drug, or 5 halflives, whichever is longer, or an unwillingness to refrain from these medications through discharge from the clinical unit. Note: Use of over-the-counter topical medications may be permitted in consultation with the Sponsor. In addition, medications for which 5 half-lives exceeds 14 days must be discussed with and approved by the Sponsor prior to subject enrollment.
16. Corticosteroid use (systemic or extensive topical) within 3 months prior to dosing.
17. Positive drug or alcohol test result or a history of alcoholism or drug abuse within 2 years prior to the first dose of study drug as defined by the Diagnostic and Statistical Manual (DSM) of Mental Disorders, 4th Edition: DSM-IV.
18. Typical consumption of ≥14 alcoholic drinks weekly. Note: 1 drink of alcohol is equivalent to ½ pint of beer (285 mL), 1 glass of spirits (25 mL), or 1 glass of wine (125 mL).
19. History of or evidence of illicit drug use within the past 2 years.
20. Surgical procedures within 4 weeks of check-in or planned elective surgery during the study period.
21. Any illness during the 4 weeks before check-in, unless deemed not clinically significant by the Investigator.
22. Known allergy to any ingredient of the study drug. Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens).
23. Inadequate venous access.
24. Currently undergoing treatment with weight loss medication or prior weight loss surgery (e.g., gastric bypass surgery).
25. Pregnant, breastfeeding, or planning to become pregnant during the study.
26. Considered by the Investigator, after reviewing medical and psychiatric history, physical examination, and laboratory evaluation, to be unsuitable for any other reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events following single oral doses of CIN-107 tablet and oral solution. | 0 to 23 days after dosing
  The safety and tolerability of CIN-107 will be assessed throughout the study based on quantitation of adverse events that occur following oral doses of CIN-107 tablet and oral solution.
Maximum concentration [Cmax] following administration of a tablet formulation of CIN-107 compared to Cmax following administration of the oral solution. | 0 to 21 days after dosing
  Cmax will be determined for CIN-107 and any other measured metabolites for participants given each formulation of baxdrostat; relative bioavailability will be evaluated by comparing these parameters between patients given the solution versus the tablet.
Cmax of CIN-107 following administration of the tablet formulation under fed versus fasted conditions. | 0 to 21 days after dosing
  Cmax will be determined for CIN-107 and any other measured metabolites for participants given baxdrostat under fed versus fasted conditions; food effect will be evaluated by comparing Cmax between participants under each condition.
Area under the curve [AUC] following administration of a tablet formulation of CIN-107 compared to AUC following administration of the oral solution. | 0 to 21 days after dosing
  Area under the curve (AUC)0-∞ and AUC0-last will be determined for baxdrostat and any other measured metabolites for participants given each formulation of baxdrostat. Then relative bioavailability will be evaluated by comparing these AUC parameters between patients given the solution versus the tablet.
Time to maximum concentration [Tmax] of CIN-107 following administration of the tablet formulation under fed versus fasted conditions. | 0 to 21 days after dosing
  Tmax will be determined for CIN-107 and any other measured metabolites for participants given baxdrostat under fed versus fasted conditions, and then food effect will be evaluated by comparing Tmax between participants under each condition.
AUC of CIN-107 following administration of the tablet formulation under fed versus fasted conditions. | 0 to 21 days after dosing
  Area under the curve (AUC)0-∞ and AUC0-last will be determined for CIN-107 and any other measured metabolites for participants given baxdrostat under fed versus fasted conditions, and then food effect will be evaluated by comparing AUC between participants under each condition.
Tmax following administration of a tablet formulation of CIN-107 compared to Tmax following administration of the oral solution. | 0 to 21 days after dosing
  Tmax will be determined for CIN-107 and any other measured metabolites for participants given each formulation of baxdrostat.

SECONDARY OUTCOMES:
Angiotensin converting enzyme (ACE) levels following single doses of CIN-107. | 0 to 21 days after dosing
  An exploratory assessment of the effect of CIN-107 on various measures associated with the Renin-Angiotensin-Aldosterone system including, but not limited to, angiotensin converting enzyme (ACE).

CONTACTS AND LOCATIONS:
Overall Officials: L Vrishabhendra, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-112&attachmentIdentifier=987d2c9f-2754-478e-bc37-f0963da20509&fileName=cin-107-112-report-synopsis_Redacted.pdf&versionIdentifier=